CLINICAL TRIAL: NCT03233295
Title: A Prospective, Single-centre, Open-label Study to Confirm the Efficacy and Safety of Vitamin D3 B.O.N. Intramuscular Injection in Adults With Vitamin D Deficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kwang Dong Pharmaceutical co., ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KDBON-CPI-01
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D deficiency (Experimental)
  Interventions: Drug: Vitamin D3 B.O.N. Injection

INTERVENTIONS:
Drug: Vitamin D3 B.O.N. Injection — cholecalciferol 200,000IU

SUMMARY:
A Prospective, Single-centre, Open-label Study to Confirm the Efficacy and Safety of Vitamin D3 B.O.N. Intramuscular Injection in adults with Vitamin D Deficiency

ELIGIBILITY:
Inclusion Criteria:

* Subjects with vitamin D deficiency

Exclusion Criteria:

* Subjects who experienced a hypersensitivity to the cholecalciferol
* Subjects with Hypercalcemia
* Subjects with Hypercalciuria
* Subjects with renal impairment
* Subjects with calcium stone
* Subjects diagnosed with sarcoidosis or pseudo-hypoparathyroidism
* Subjects who are to take vitamin D supplements during the study period

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2016-08-27 (Actual); Study Completion 2016-08-27 (Actual)

PRIMARY OUTCOMES:
serum 25(OH)D concentration | 12 months

SECONDARY OUTCOMES:
serum 1,25(OH)2D concentration | 12 months

IPD SHARING:
Plan to Share IPD: No